CLINICAL TRIAL: NCT03561805
Title: Prolonged Continuous ECG Monitoring Prior to TrAnscatheter AoRtic ValvE Implantation: the PARE Study
Brief Title: Prolonged Continuous ECG Monitoring Prior to Transcatheter Aortic Valve Implantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal investigator, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARE
Record Dates: First submitted 2018-04-13; First posted 2018-06-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-06

CONDITIONS: Aortic Valve Stenosis; Arrythmia
Keywords: TAVI; ECG monitoring
MeSH Terms: conditions — Aortic Valve Stenosis; Arrhythmias, Cardiac | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prolonged continuous ECG monitoring (Other): Patients will undergo a prolonged continuous ECG monitoring using the CardioSTAT® device within the 3 months prior to the TAVI procedure. The duration of the ECG monitoring will be of 1 week.
  Interventions: Device: ECG monitoring

INTERVENTIONS:
Device: ECG monitoring — Prolonged continuous ECG monitoring using the CardioSTAT® device within the 3 months prior to the TAVI procedure

SUMMARY:
Patients with severe aortic stenosis candidates for a TAVI procedure harbor a high burden of silent arrhythmic events. Pre-procedural detection of such arrhythmias should help the investigators to implement specific therapeutic measures that may improve patient outcomes and reduce hospitalization length post-TAVI.

DETAILED DESCRIPTION:
This is a prospective registry including patients accepted by the heart team for a TAVI procedure. Patients will undergo a prolonged continuous ECG monitoring using the CardioSTAT® device within the 3 months prior to the TAVI procedure. The duration of the ECG monitoring will be of 1 week. There will be no restriction regarding the type of valve and approach used for the TAVI procedure. All type of arrhythmic events will be recorded, as well as the specific therapeutic measures implemented upon the occurrence of the arrhythmic event. Following the TAVI procedure, the patients will be monitored (telemetry) until hospital discharge. All arrhythmic events during the hospitalization period will be recorded. Clinical follow-up will be performed at 30 days, and 1 year post-TAVI, and yearly thereafter up to 5-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe aortic stenosis accepted for a TAVI procedure by the Heart Team.

Exclusion Criteria:

* Urgent TAVI procedure or logistic reasons precluding an ECG monitoring of at least 1 week within the 3 months prior to the TAVI procedure.
* Prior permanent pacemaker.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Arrhythmic events | Within 3 months prior to the TAVI procedure
  Incidence and type of arrhythmic events
Therapeutic changes | Within 3 months prior to the TAVI procedure
  incidence of arrhythmic events identified by the device leading to therapeutic changes prior to the TAVI procedure

SECONDARY OUTCOMES:
Atrial fibrillation | Within 3 months prior to the TAVI procedure
  incidence of atrial fibrillation
Atrial fibrillation | Within 3 months prior to the TAVI procedure
  duration of atrial fibrillation
Atrioventricular block | Within 3 months prior to the TAVI procedure
  incidence of advanced atrioventricular block
Severe bradycardia | Within 3 months prior to the TAVI procedure
  incidence of severe bradycardia
Left bundle branch block | Within 3 months prior to the TAVI procedure
  incidence of left bundle branch block
Permanent pacemaker | Within 3 months prior to the TAVI procedure
  percentage of patients with an indication of permanent pacemaker
Anticoagulation therapy | Within 3 months prior to the TAVI procedure
  percentage of patients with an indication for anticoagulation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No